CLINICAL TRIAL: NCT04950569
Title: Levosimendan Improves Heart Failure Through Regulating 3 Cardiac Specific miRNAs (miR-660-3p, miR-665 and miR-1285-3p) in Patients With Refractory Heart Failure (NYHA III-IV)
Brief Title: Effect of Levosimendan on miRNAs Regulation in the Failing Hearts
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Li Ni, Associate Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJ-LS-HF
Record Dates: First submitted 2021-06-24; First posted 2021-07-06 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: Heart Failure; Levosimendan; MicroRNA
MeSH Terms: conditions — Heart Failure | interventions — Simendan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levosimendan (Experimental): Receive standard heart failure treatment, plus levosimendan treatment.
  Interventions: Drug: levosimendan
- Control (No Intervention): Receive standard heart failure treatment, without levosimendan treatment.

INTERVENTIONS:
Drug: levosimendan — On the basis of standard conventional anti-heart failure treatment, levosimendan was used for 24 hours. The first load was 12 μg/kg, intravenous injection for 10 minutes, followed by intravenous infusion of 0.1 μg/Kg/min for 24 hours.
  Arms: Levosimendan

SUMMARY:
Chronic heart failure is the terminal stage of various cardiovascular diseases. It is characterized with high fatality rate and high recurrence rate, which brings a heavy economic burden to patients and society. Although in recent years, the long-term prognosis of patients with heart failure has been greatly improved by the advances in drugs and new techniques, some patients have eventually progressed to refractory heart failure.

The newly developed positive inotropic drug levosimendan is a new type of calcium sensitizer, increasing the sensitivity of troponin to calcium ions, without directly increasing the concentration of calcium ions in cardiomyocytes. Levosimendan improves heart function by increasing myocardial contractility, dilating blood vessels, regulating coronary blood flow, and also exhibits anti-inflammatory, anti-oxidant and anti-apoptotic effects. Compared with traditional inotropic drugs, levosimendan does not increase calcium ion concentration or increase oxygen consumption. And it does not easily lead to malignant arrhythmia or increase the long-term mortality of patients. Because of its long half-life, intermittent use of levosimendan can improve contractile function for a long time, thereby effectively alleviating the symptoms of patients with advanced heart failure. Patients treated with levosimendan had a higher survival rate, fewer hospitalizations, and a greatly improved quality of life.

MicroRNAs (miRNAs) are a class of non-coding RNAs with important regulatory roles. They are 22-nucleotide single-stranded RNAs derived from endogenous hairpin structure transcripts. MiRNAs are reported to be involved in the pathological process of heart remodeling. MiRNAs can be secreted by cells into the peripheral blood and exist stably, which can be used as new diagnostic markers for various diseases. The investigators have previously conducted simultaneous detection of miRNAs in myocardial tissue and peripheral blood in patients with heart failure, and conducted an epidemiological follow-up study. The investigators have identified three cardiac-specific secretory miRNAs (miR-660-3p, miR-665 and miR-1285-3p) which are significantly up-regulated in the plasma of patients with chronic heart failure. Subsequent analysis proved them as valuable biomarkers for the diagnosis and prognosis of heart failure.

The investigators hypothesis that the new positive inotropic drug levosimendan improve heart function by regulating the miRNAs in patients with heart failure. This study aims to treat patients with advanced heart failure with levosimendan. By combining the expression of myocardial specific miRNAs, myocardial injury markers, hemodynamics, patient symptoms, long-term prognosis and other clinical indicators, the investigators will explore the relationship between the three myocardial-specific miRNAs expression and cardiac function improvement by levosimendan treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age over 18 years old, no gender limit;
2. A clear diagnosis of chronic systolic heart failure with heart function NYHA III-IV (including medical history, clinical symptoms, and signs) by two attending physicians or above the level of attending ;
3. Left ventricular ejection fraction (LVEF) <40%;
4. Plasma NT-proBNP>1000 ng/L;
5. Participate voluntarily and sign an informed consent form, and can be followed up for more than 6 months.

Exclusion Criteria:

1. NYHA Class I-II of cardiac function;
2. Acute myocardial infarction occurred in the past month;
3. Unstable angina pectoris;
4. Patients with acute pulmonary edema or acute hemodynamic disturbance;
5. Right heart failure due to lung disease;
6. Patients who are going to undergo heart transplantation or cardiac resynchronization therapy (CRT), or those who have received CRT treatment;
7. Female patients who have or plan to become pregnant;
8. Those who have participated in any drug clinical trials within the previous 3 months;
9. Those who have a history of tumors or are currently suffering from tumors, or pathological examinations have confirmed precancerous lesions (such as ductal carcinoma in situ of the breast, or dysplasia of the cervix);
10. Patients who was detected with a malignant mass in the body through examination (physical examination, or X-ray examination or B-ultrasound examination or other means), or detected with a hyperplastic gland or adenoma that has endocrine activity and affects heart function or endocrine function, such as pheochromocytoma, etc.;
11. The patient refused to comply with the requirements of this research to complete the research work;
12. According to the judgment of the investigator, the patient cannot complete the study or cannot comply with the requirements of the study (due to management reasons or other reasons).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2020-10-29 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP | From the day before levosimendan treatment to the 7th day after levosimendan treatment.
  Change of blood N-terminal prohormone of brain natriuretic peptide (NT-proBNP) level in 7 days

SECONDARY OUTCOMES:
miR-660-3p, miR-665 and miR-1285-3p | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Levels of the 3 cardiac specific miRNAs (miR-660-3p, miR-665 and miR-1285-3p) in blood, denoted as the fold change of the miRNA (miR-660-3p, miR-665 and miR-1285-3p) read copies over the the mRNA read copy of U6 promoter (loading control).
Left ventricular ejection fraction | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Left ventricular ejection fraction by echocardiography to evaluate cardiac function
NYHA | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Assessment of cardiac function by New York Heart Association (NYHA) classification. Cardiac function is assessed from Class I to Class IV by NYHA. Higher class indicates worse cardiac function.
6 minutes walking distance | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Assessment of cardiac function by 6 minutes walking distance

OTHER OUTCOMES:
Occurrence of cardiovascular death or heart transplant | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Death owing to cardiovascular reasons or heart transplant
Occurrence of all-cause death | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Death owing to all causes
Frequency of recurrent exacerbation of heart failure | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Frequency of recurrent exacerbation of heart failure symptoms
Frequency of re-hospitalization for cardiovascular reasons | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Frequency of re-hospitalization for cardiovascular reasons
Score by the Minnesota Quality of Life Scale | From the day before levosimendan treatment to the 6th month after levosimendan treatment.
  Assessment of quality of life by Minnesota Quality of Life Scale for heart condition. The score ranges from 0 to 105. Higher score represents worse heart condition.

CONTACTS AND LOCATIONS:
Overall Officials: Li Ni, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No